CLINICAL TRIAL: NCT07267741
Title: The Impact of Using Virtual Reality Technology on Depression, Anxiety, and Stress Among Palestinian Patients Undergoing Breast Biopsy: Randomized Controlled Trial
Brief Title: Using Virtual Reality Technology on Depression, Anxiety, and Stress Among Palestinian Patients Undergoing Breast Biopsy
Acronym: VR/RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nablus University for Vocational and Technical Education (Other)
Responsible Party: Principal Investigator, Khulood Mansour, Principal Investigator, Nablus University for Vocational and Technical Education
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Nrs.September2025/6
Record Dates: First submitted 2025-11-18; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-10

CONDITIONS: Depression; Anxiety; Stress
Keywords: Virtual Reality Technology; Depression; Anxiety; Stress; Breast Biopsy; Palestinian Patients
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants in the VR group will wear a VR headset, while the control group will receive standard care without VR. The intervention involves a VR application featuring immersive 360-degree natural environments, including peaceful forests, tranquil beaches, and serene gardens. Patients can choose one environment, enhanced by relaxing music and nature sounds. VR sessions will last 15 to 30 minutes, with the headset used to immerse patients in their selected calming environment. The session will be terminated if the patient experiences discomfort or requests removal.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR group (Experimental): The VR group will utilize a head-mounted VR headset with built-in headphones. Patients will be selected for VR environments from a predefined list of natural scenes. VR will be applied during the procedure, with sessions lasting 15 to 30 minutes.
  Interventions: Device: Meta Quest 2 VR headset
- control group (No Intervention): Participants will receive only standard care according to the hospital protocol during the procedure.

INTERVENTIONS:
Device: Meta Quest 2 VR headset — The VR intervention will utilize a head-mounted VR headset with built-in headphones. Patients will be selected for VR environments from a predefined list of natural scenes, including a tropical beach, diving, forest, and snowy landscape, each accompanied by relaxing music and nature sounds. The Guided Meditation VR application from Cubicle Ninjas (https://guidedmeditationvr.com/) provides 360-degree immersive nature environments with standardized calming background audio. VR will be applied during the procedure, with sessions lasting 15 to 30 minutes and discontinued if the patient experiences nausea, dizziness, or requests removal.
  Arms: VR group

SUMMARY:
The goal of this randomized controlled trial was to investigate the impact of Virtual Reality (VR) technology on depression, anxiety, and stress levels among Palestinian patients undergoing breast biopsy. The study aimed to evaluate the effectiveness of VR as a non-pharmacological intervention to reduce psychological distress associated with the biopsy procedure.

The main research hypotheses are:

H01: There will be no significant difference in depression levels between patients who receive immersive VR during breast biopsy and those who receive standard care.

H02: There will be no significant difference in anxiety levels between patients who receive immersive VR during breast biopsy and those who receive standard care.

H03: There will be no significant difference in stress levels between patients who receive immersive VR during breast biopsy and those who receive standard care.

Participants will:

Receive either a VR intervention or standard care during their breast biopsy. Wear a VR headset for 15-30 minutes, experiencing a calming virtual environment designed to promote relaxation.

Complete assessments of depression, anxiety, and stress before and after the procedure using validated psychological questionnaires.

DETAILED DESCRIPTION:
Title: The Impact of Using Virtual Reality Technology on Depression, Anxiety, and Stress Among Palestinian Patients Undergoing Breast Biopsy: A Randomized Controlled Trial

Background:

Breast biopsy is an essential diagnostic procedure for detecting breast abnormalities but often induces significant psychological distress, including depression, anxiety, and stress, which can negatively affect patient wellbeing and procedure outcomes. Virtual Reality (VR) technology provides immersive and calming environments that may help alleviate these emotional burdens without pharmacological intervention. This study aims to assess the effectiveness of VR in reducing depression, anxiety, and stress among Palestinian patients undergoing breast biopsy.

Methods:

A randomized controlled trial will be conducted at a healthcare facility in Palestine, enrolling a total of 80 patients scheduled for breast biopsy. Participants will be randomly assigned to either the VR intervention group (n=40) or the control group receiving standard care (n=40). The VR group will wear a head-mounted VR device for 15 to 30 minutes during the biopsy, immersing themselves in soothing virtual environments such as peaceful natural landscapes with accompanying relaxing music and nature sounds. Psychological assessments measuring depression, anxiety, and stress levels will be administered before and after the procedure using validated questionnaires. The data collection and intervention period will span approximately two months.

ELIGIBILITY:
Inclusion Criteria:

* Female patients scheduled to undergo a breast biopsy.
* Patients older than 18 years.
* Patients who are able to provide informed consent.
* Patients with no prior history of severe psychiatric disorders that could affect the assessment of depression, anxiety, or stress.
* Patients who are willing and able to participate in the VR intervention and complete self-report questionnaires.

Exclusion Criteria:

* Patients who have a history of severe psychiatric disorders, epilepsy, hypertension, or chronic pain.
* Patients who are mute and cannot read or write, patients with visual, hearing, or cognitive impairment.
* Patients who have implanted hearing aids or cardiac pacemakers.
* Patients who will receive any anxiolytic, sedative, or hypnotic drugs before or during the procedure.
* Patients who may be exposed to complications during the procedure.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2026-01-10 (Estimated); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
Depression Anxiety Stress Scale-21 (DASS21) | before the procedure and then 60 minutes post-procedure
  (DASS21) consists of 21 statements designed to measure symptoms of depression, anxiety, and stress experienced over the past week. Each statement is rated on a 4-point scale from 0 to 3.

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) cannot be shared due to ethical concerns about participant privacy and the inappropriate use of data. Also, compliance with journal publication policies

REFERENCES:
- See also: the website Guided Meditation VR application, developed by Cubicle Ninjas Agency — https://guidedmeditationvr.com/